CLINICAL TRIAL: NCT06721507
Title: Preoperative Tirzepatide for Bariatric Surgery
Brief Title: 2024 Tirzepatide-Bariatric Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Marlene Starr (Other)
Responsible Party: Sponsor-Investigator, Marlene Starr, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 97933
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Obesity and Obesity-related Medical Conditions; Bariatric Surgery
MeSH Terms: conditions — Obesity | interventions — Tirzepatide; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care plus Drug (Experimental): Participant receives drug for 3 months prior to surgery
  Interventions: Drug: tirzepatide
- Standard of Care Alone (Active Comparator)
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Drug: tirzepatide — Participants will be educated on dietary and lifestyle changes. Participants will self inject 2.5 mg tirzepatide subcutaneously once weekly and maintain a drug administration diary. Dose escalation will proceed per package directions if instructed by study team at follow up visits.
  Other Names: Mounjaro; Zepbound
  Arms: Standard of Care plus Drug
Behavioral: Standard of Care — Participants will be educated on dietary and lifestyle changes
  Arms: Standard of Care Alone

SUMMARY:
This clinical trial will test whether preoperative tirzepatide treatment improves outcomes after bariatric surgery. The outcome of this study could impact therapeutic guidelines for the multimodal treatment of obesity.

The major objectives are:

1. To evaluate whether pre-operative tirzepatide treatment reduces tissue and circulating inflammatory markers at the time of surgery.
2. To establish the relationship of these changes with postoperative improvements in weight loss, metabolic and inflammatory profiles, comorbidity resolution (glycemic control, blood pressure, lipid profile), and 30-day surgical complications. Researchers will compare data from patients taking tirzepatide to data from patients not taking tirzepatide before their planned bariatric surgery to see if tirzepatide reduces inflammation and improves health outcomes after bariatric surgery.

Participants will:

Take or not take tirzepatide, depending on what study group they are in, once a week for 3 months.

Visit the endocrine clinic once a month for 3 months to be prescribed the drug and for checkups regarding side effects due to the drug.

Keep a diary to document taking the drug and any side effects. Continue with their planned bariatric surgery and post-surgery follow-ups according to their healthcare provider.

ELIGIBILITY:
Inclusion Criteria:

* adults who have been enrolled in the multidisciplinary metabolic and bariatric surgery program at the UK HealthCare Weight Loss Surgery Clinic and are scheduled to receive laparoscopic or robotic sleeve gastrectomy, or gastric bypass surgery
* BMI greater than or equal to 40 kg/m2 with one or more obesity-related comorbidities
* have demonstrated abstinence from any form of nicotine use, confirmed by serum nicotine and metabolite testing
* enrollment in the ADORE Bariatric Tissue Bank (IRB #69767)

Exclusion Criteria:

* any contraindication to the use of tirzepatide (per package insert)
* Personal or family history of medullary thyroid carcinoma
* Patients with Multiple Endocrine Neoplasm syndrome type 2
* Hypersensitivity to tirzepatide
* History of pancreatitis
* Type 1 Diabetes
* patients with active, untreated or symptomatic cholelithiasis or jaundice
* consistent use of a GLP-1 or GLP-1/GIP receptor agonist, over the past 90 days
* diagnosed autoimmune disease
* current use of immunosuppressive agents or use within the past 30 days
* moderate or severe substance use disorder according to DSM-5 criteria
* uncontrolled significant psychiatric disorder as assessed by specialized bariatric psychologist
* female participant who is pregnant, breast-feeding, or intends to become pregnant with in 1 year following surgery
* a prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in inflammatory markers c reactive protein (CRP) | Baseline and 3 months post-drug
  Inflammatory marker will be measured by ELISA in blood samples drawn from patient.
Change in inflammatory markers interleukin 6 (IL-6) | Baseline and 3 months post-drug
  Inflammatory marker will be measured by ELISA in blood samples drawn from patient.
Change in inflammatory markers tumor necrosis factor (TNF) | Baseline and 3 months post-drug
  Inflammatory marker will be measured by ELISA in blood samples drawn from patient.
change in inflammatory markers (leptin) | Baseline and 3 months post-drug
  Inflammatory marker will be measured by ELISA in blood samples drawn from patient.
change in inflammatory markers (adiponectin) | Baseline and 3 months post-drug
  Inflammatory marker will be measured by ELISA in blood samples drawn from patient.
change in inflammatory markers renin-angiotensin-aldosterone system (RAAS) | Baseline and 3 months post-drug
  Inflammatory markers will be measured by ELISA in blood samples drawn from patient.
RNA sequencing | at time of surgery
  Bulk RNA sequencing analyses will be performed on tissue samples of fat and liver collected at the time of surgery

SECONDARY OUTCOMES:
Change in weight | Baseline, 3 months post-drug, 1-, 3-, 6-, and 12-months post surgery
  patient weight will be measured
30-day surgical complications | 1-, 3-, 6-, and 12-months post surgery
  Surgical complications will be assessed as standard of care and data evaluated for this study
change in inflammatory markers c reactive protein (CRP) | 1-, 3-, 6-, and 12-months post surgery
  Inflammatory marker will be measured by ELISA in blood samples drawn from patient.
change in inflammatory markers interleukin 6 (IL-6) | 1-, 3-, 6-, and 12-months post surgery
  Inflammatory marker will be measured by ELISA in blood samples drawn from patient.
change in inflammatory markers tumor necrosis factor (TNF) | 1-, 3-, 6-, and 12-months post surgery
  Inflammatory marker will be measured by ELISA in blood samples drawn from patient.
change in inflammatory markers (leptin) | 1-, 3-, 6-, and 12-months post surgery
  Inflammatory marker will be measured by ELISA in blood samples drawn from patient.
change in inflammatory markers (adiponectin) | 1-, 3-, 6-, and 12-months post surgery
  Inflammatory marker will be measured by ELISA in blood samples drawn from patient.
change in inflammatory markers renin-angiotensin-aldosterone system (RAAS) | 1-, 3-, 6-, and 12-months post surgery
  Inflammatory marker will be measured by ELISA in blood samples drawn from patient.
change in blood pressure | Baseline, 3 months post-drug, 1-, 3-, 6-, and 12-months post surgery
  blood pressure per standard method in clinic
Change in Hemoglobin A1c | Baseline, 3 months post-drug, 1-, 3-, 6-, and 12-months post surgery
  HbA1c will be measured by clinic lab
change in blood glucose | Baseline, 3 months post-drug, 1-, 3-, 6-, and 12-months post surgery
  blood glucose will me measured in clinic lab
change in cholesterol | Baseline, 3 months post-drug, 1-, 3-, 6-, and 12-months post surgery
  cholesterol measured in clinic lab
change in high-density lipoprotein (HDL) | Baseline, 3 months post-drug, 1-, 3-, 6-, and 12-months post surgery
  high-density lipoprotein (HDL) measured in clinic lab
change in low-density lipoprotein (LDL) | Baseline, 3 months post-drug, 1-, 3-, 6-, and 12-months post surgery
  low-density lipoprotein measured by clinic lab
change in triglycerides | Baseline, 3 months post-drug, 1-, 3-, 6-, and 12-months post surgery
  triglycerides measured in clinic lab
change in insulin | Baseline, 3 months, post-drug, 1-, 6-, and 12-months post surgery
  insulin measured in clinic lab

CONTACTS AND LOCATIONS:
Overall Officials: Marlene Starr, PhD, Principal Investigator — University of Kentucky; Varun Jain, MD, Study Director — University of Kentucky; William B Inabnet, MD, Study Director — University of Kentucky; Simon J Fisher, MD. PhD, Study Director — University of Kentucky; Philip A Kern, MD, Study Director — University of Kentucky; Barbara Nikolajczyk, PhD, Study Director — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No